CLINICAL TRIAL: NCT06531850
Title: Prospective Study of Serum Marker LncRNA RP5-977B1 for Differentiating Benign
Brief Title: Prospective Study of Serum Marker LncRNA RP5-977B1 in Pulmonary Nodules
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2023-013(JYK)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-01

CONDITIONS: Tumor of Lung; Pulmonary Nodule
Keywords: lung cancer; RP5-977B1; LncRNA
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign nodule: * Pulmonary nodules were detected by imaging and surgically resected.
    * Age 15-75 years old.
      * Surgery or puncture is to be performed for pathological diagnosis. ④ Adequate hematological function and liver and kidney function reserve. ⑤ The sample has no hemolysis, sufficient margin, and the source record is clear and can be checked.
- Tumor: * Pulmonary nodules were detected by imaging and surgically resected.
    * Age 15-75 years old.
      * Surgery or puncture is to be performed for pathological diagnosis. ④ Adequate hematological function and liver and kidney function reserve. ⑤ The sample has no hemolysis, sufficient margin, and the source record is clear and can be checked.

SUMMARY:
Based on previous studies, this project intends to use prospective studies to select patients identified by imaging as pulmonary nodules to explore the potential of RP5-977B1 in differentiating benign and malignant pulmonary nodules, construct diagnostic models combined with clinical protein tumor markers, compare the diagnostic efficacy of the two, and finally determine the sensitivity and specificity of markers through pathological results. It provides a new content for the diagnosis of benign and malignant pulmonary nodules.

DETAILED DESCRIPTION:
For the purpose of clinical diagnosis, disease monitoring, treatment or prognosis assessment, patients with pulmonary nodules may need to draw blood for routine laboratory tests several times during diagnosis and treatment. There may be some blood samples to be discarded after the completion of routine tests. This clinical trial will only use these remaining blood samples as research samples. The samples collected in this part of the study were serum samples from patients with pulmonary nodules, and 50 subjects were planned to be enrolled.

Admission criteria: ① Pulmonary nodules were detected by imaging and surgically resected.

② Age 15-75 years old.

* Surgery or puncture is to be performed for pathological diagnosis.

  * Adequate hematological function and liver and kidney function reserve. ⑤ The sample has no hemolysis, sufficient margin, and the source record is clear and can be checked.

Exclusion criteria: ① Patient samples have hemolysis, have been contaminated, have been placed for too long, have insufficient sample allowance, and have mixed records.

* History of malignant tumor.

  * Serious underlying diseases and complications may affect systemic treatment. ④ Can not guarantee to receive blood tests on time.

    * Received anti-tumor Chinese medicine, immunization, chemotherapy and other treatments within 2 weeks.

Exclusion criteria: ① Subjects who do not meet the inclusion criteria or who meet the exclusion criteria and are mistakenly enrolled.

* Samples collected for two or more times from the same patient should be retained only the samples collected for the first time, and all subsequent samples collected should be excluded.

  * Samples with incomplete case information. ④ Sample quality control unqualified samples due to sample collection, storage, transportation and other reasons.

    * Samples that cannot be tested due to instruments and other reasons.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary nodules were detected by imaging and surgically resected.

  * Age 15-75 years old.

    * Surgery or puncture is to be performed for pathological diagnosis.

      * Adequate hematological function and liver and kidney function reserve. ⑤ The sample has no hemolysis, sufficient margin, and the source record is clear and can be checked.

Exclusion Criteria:

* Patient samples have hemolysis, have been contaminated, have been placed for too long, have insufficient sample allowance, and record mixed samples.

  * History of malignant tumor. ③ Serious underlying diseases and complications may affect systemic treatment. ④ Can not guarantee to receive blood tests on time. ⑤ Received anti-tumor Chinese medicine, immunization, chemotherapy and other treatments within 2 weeks.

Ages: 15 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Serum samples from patients with radiographic findings and surgical removal of pulmonary nodules were selected.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Benign nodule | A week
  Pathological findings determined that the nodules were benign in the patient
Tumor | A week
  Pathological findings identified the nodules as malignant tumors in the patient

CONTACTS AND LOCATIONS:
Overall Officials: Zijian Wu, Learned, Study Chair — Cancer Hospital & Affiliated Guangzhou Medical University
Locations (1):
- Cancer Hospital & Affiliated Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Due to the requirements of the institution and the need to protect the privacy of patients, it is not convenient to disclose IPD.